CLINICAL TRIAL: NCT01083316
Title: Phase II Trial of Induction Therapy With Bortezomib and Dexamethasone Followed by High-Dose Melphalan and Stem Cell Transplantation in Patients With AL Amyloidosis
Brief Title: Bortezomib and Dexamethasone Followed by High-Dose Melphalan and Stem Cell Transplantation for Primary (AL) Amyloidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-28441; X05292 (Other: Millennium)
Record Dates: First submitted 2009-11-02; First posted 2010-03-09 (Estimated); Results first posted 2017-02-06 (Estimated); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Amyloidosis
Keywords: Amyloid; Amyloidosis; AL Amyloidosis; Primary Amyloidosis; Stem Cell Transplant
MeSH Terms: conditions — Amyloidosis; Alzheimer Disease; Immunoglobulin Light-chain Amyloidosis | interventions — Bortezomib; Dexamethasone; Calcium Dobesilate; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single Arm - Investigational (Experimental): Induction:
  Bortezomib (Velcade) 1.3 mg/m2/dose IV Days 1, 4, 8, 11 repeated every 21 days
  Dexamethasone 20 mg PO/IV Days 1, 4, 8, 11 repeated every 21 days
  Conditioning:
  Bortezomib 1.0 mg/m2/dose will be administered on Days +6, -3, +1, + 4
  Melphalan 70-100 mg/m2/day IV on days -2 and -1
  Interventions: Drug: Bortezomib; Drug: Dexamethasone; Drug: Melphalan

INTERVENTIONS:
Drug: Bortezomib — Induction:
  Velcade 1.3 mg/m2/dose IV Days 1, 4, 8, 11 repeated every 21 days
  Conditioning:
  Bortezomib 1.0 mg/m2/dose will be administered on Days +6, -3, +1, + 4
  Other Names: Velcade
Drug: Dexamethasone — Induction:
  Dexamethasone 20 mg PO/IV Days 1, 4, 8, 11 repeated every 21 days
  Other Names: Decadron
Drug: Melphalan — Conditioning:
  Melphalan 70-100 mg/m2/day IV on days -2 and -1
  Other Names: Alkeran

SUMMARY:
The drugs dexamethasone and bortezomib are both FDA-approved for the treatment of multiple myeloma, a disease very similar to amyloidosis. However, they are currently investigational for the treatment of amyloidosis.

We want to find out if the addition of dexamethasone and bortezomib to standard high dose chemotherapy and stem cell transplant can help improve response.

Standard treatment includes four steps: 1) Stem Cell Mobilization (standard) 2) Stem Cell Collection (standard) 3) Conditioning Regimen (Melphalan chemotherapy). The conditioning regimen helps to kill the abnormal cells in the body and makes room in the bone marrow for new blood stem cells to grow. 4) Stem Cell Infusion

Participants in this study will have an additional treatment step called "induction therapy", designed as the first step towards reducing the number of abnormal cells in the body. Two cycles of the investigational drugs bortezomib and dexamethasone will be given during induction therapy. In addition, bortezomib will given as part of the conditioning regimen, in addition to the standard melphalan chemotherapy.

DETAILED DESCRIPTION:
The drugs dexamethasone and bortezomib are both FDA-approved drugs for the treatment of multiple myeloma, a disease very similar to amyloidosis. However, they are currently investigational for the treatment of amyloidosis.

The investigators want to find out if the addition of dexamethasone and bortezomib to standard treatment of high dose chemotherapy and stem cell transplant can help improve response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of primary systemic (AL) amyloidosis based on:

  1. Deposition of amyloid material by congo red stain showing characteristic green birefringence, and
  2. monoclonal light chain protein in the serum or urine or immunohistochemical studies or serum free light chain assay and
  3. evidence of tissue involvement other than carpal tunnel syndrome, i.e. positive immunohistochemical staining of bone marrow demonstrating clonal plasma cells; or tissue amyloid deposits with anti-kappa or anti-lambda anti-serum; evidence for a plasma cell dyscrasia (PCD) by serum/urine or bone marrow; or overwhelmingly convincing clinical features e.g. macroglossia, associated with other systemic manifestations.

     Note: Patients with senile, secondary, localized, dialysis-related or familial amyloidosis are not eligible. Confirmation of tissue diagnosis at all sites of organ dysfunction is encouraged, but not required.
* Must be at least 18 years of age.
* Must have a performance status of 0-2 by Southwest Oncology Group criteria
* Must have left ventricular ejection fraction (LVEF) at least 45% by echocardiogram within 60 days of enrollment
* Prior chemotherapy with alkylating agent allowed only if no evidence of Myelodysplastic Dysplastic Syndrome (MDS) morphologically or cytogenetically. Total cumulative dose of oral melphalan must be less than 300 mg. Patients should not have received any cytotoxic therapy less than 4 weeks prior to registration and should have fully recovered from the effects of such therapy.
* Pulmonary Function Tests must show Diffusing capacity of the lungs for carbon monoxide (DLCO) at least 50%.
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
* Male subject agrees to use an acceptable method for contraception for the duration of the study.

Exclusion Criteria:

* No overt multiple myeloma (over 30% bone marrow plasmacytosis, extensive (great than 2) lytic lesions, hypercalcemia).
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 3 years.
* No known to be HIV positive.
* No platelet count of less than or equal to 70,000 within 14 days before enrollment.
* No absolute neutrophil count of less than or equal to 1000 within 14 days before enrollment.
* No greater than or equal to Grade 2 peripheral neuropathy within 14 days before enrollment.
* No myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure (see section 8.4), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
* No hypersensitivity to bortezomib, boron or mannitol.
* No pregnant or breast-feeding females. Confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Must not have received other investigational drugs with 14 days before enrollment
* No serious medical or psychiatric illness likely to interfere with participation in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2013-08 (Actual); Study Completion 2020-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vaishali Sanchorawala, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Boston Medical Center Active Clinical Trials — http://www.bumc.bu.edu/clinicaltrials

RESULTS

PARTICIPANT FLOW:
Groups:
- Bortezomib and Dexamethasone: Induction:
  Bortezomib (Velcade) 1.3 mg/m2/dose IV Days 1, 4, 8, 11 repeated every 21 days Dexamethasone 20 mg PO/IV Days 1, 4, 8, 11 repeated every 21 days
  Conditioning:
  Bortezomib 1.0 mg/m2/dose will be administered on Days +6, -3, +1, + 4 Melphalan 70-100 mg/m2/day IV on days -2 and -1
  Bortezomib (Velcade) and Dexamethasone: Induction:
  Velcade 1.3 mg/m2/dose IV Days 1, 4, 8, 11 repeated every 21 days
  Dexamethasone 20 mg PO/IV Days 1, 4, 8, 11 repeated every 21 days
  Conditioning:
  Bortezomib 1.0 mg/m2/dose will be administered on Days +6, -3, +1, + 4
  Melphalan 70-100 mg/m2/day IV on days -2 and -1
Period: Overall Study
Arm/Group | Bortezomib and Dexamethasone
Started | 35
Completed | 32
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Bortezomib and Dexamethasone: Induction:
  Bortezomib (Velcade) 1.3 mg/m2/dose intravenous (IV) Days 1, 4, 8, 11 repeated every 21 days Dexamethasone 20 mg PO/IV Days 1, 4, 8, 11 repeated every 21 days
  Conditioning:
  Bortezomib 1.0 mg/m2/dose will be administered on Days +6, -3, +1, + 4 Melphalan 70-100 mg/m2/day IV on days -2 and -1
  Bortezomib (Velcade) and Dexamethasone: Induction:
  Velcade 1.3 mg/m2/dose IV Days 1, 4, 8, 11 repeated every 21 days
  Dexamethasone 20 mg PO/IV Days 1, 4, 8, 11 repeated every 21 days
  Conditioning:
  Bortezomib 1.0 mg/m2/dose will be administered on Days +6, -3, +1, + 4
  Melphalan 70-100 mg/m2/day IV on days -2 and -1
Arm/Group | Bortezomib and Dexamethasone
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Disease Response
Description: Complete response: Normal serum free light chain ratio and Negative serum and urine immunofixation electrophoresis Very good partial response: Difference in serum free light chains less than 40 mg/L Partial Response: >50% Reduction in the difference in serum free light chains
Time Frame: One year
Measure: Count of Participants; unit: Participants
Arm/Group | Bortezomib and Dexamethasone
Number analyzed (Participants) | 26
Participants | 20

2. Primary Outcome: Number of Participants Surviving at 100 Days Post Transplant
Time Frame: 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | Bortezomib and Dexamethasone
Number analyzed (Participants) | 30
Participants | 27

3. Primary Outcome: Number of Participants Proceeding to Transplant Following Induction
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bortezomib and Dexamethasone
Number analyzed (Participants) | 35
Participants | 30

4. Secondary Outcome: Number of Participants Surviving at 5 Years
Time Frame: 5 years
Population: number of patients that completed at least one cycle of induction therapy
Measure: Count of Participants; unit: Participants
Groups:
- Bortezomib and Dexamethasone: Induction:
  Bortezomib (Velcade) 1.3 mg/m2/dose IV Days 1, 4, 8, 11 repeated every 21 days
  Dexamethasone 20 mg PO/IV Days 1, 4, 8, 11 repeated every 21 days
  Conditioning:
  Bortezomib 1.0 mg/m2/dose will be administered on Days +6, -3, +1, + 4
  Melphalan 70-100 mg/m2/day IV on days -2 and -1
  Bortezomib: Induction:
  Velcade 1.3 mg/m2/dose IV Days 1, 4, 8, 11 repeated every 21 days
  Conditioning:
  Bortezomib 1.0 mg/m2/dose will be administered on Days +6, -3, +1, + 4
  Dexamethasone: Induction:
  Dexamethasone 20 mg PO/IV Days 1, 4, 8, 11 repeated every 21 days
  Melphalan: Conditioning:
  Melphalan 70-100 mg/m2/day IV on days -2 and -1
Arm/Group | Bortezomib and Dexamethasone
Number analyzed (Participants) | 35
Participants | 29

ADVERSE EVENTS:
Time Frame: 100 days
Arm/Group | Bortezomib and Dexamethasone
Serious Adverse Events (participants affected / at risk) | 35/35
Other Adverse Events (participants affected / at risk) | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortezomib and Dexamethasone (N=35)
autograft versus host disease (Immune system disorders) | 2 (2)
neutropenic fever (Blood and lymphatic system disorders) | 7 (7)
fever (General disorders) | 7
Acute kidney failure (Renal and urinary disorders) | 3 (3)
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
cardiac arrest (Cardiac disorders) | 1 (1)
creatinine increased (Investigations) | 1 (1)
diarrhea (Gastrointestinal disorders) | 15 (15)
Epstein Barr Virus-related Polymorphous Post Transplant Lymphoproliferative disorder (Blood and lymphatic system disorders) | 1 (1)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
fatigue (General disorders) | 18 (18)
gastrointestinal bleed (Gastrointestinal disorders) | 1 (1)
hemorrhoidal hemmorhage (Gastrointestinal disorders) | 1 (1)
invasive aspirgillosis (Infections and infestations) | 1 (1)
multiorgan failure (General disorders) | 1 (1)
nausea (General disorders) | 6 (6)
sepsis (Infections and infestations) | 4 (4)
syncope (Nervous system disorders) | 8 (9)
thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
stomatitis (Infections and infestations) | 1 (1)
skin rash (Skin and subcutaneous tissue disorders) | 3 (3)
hypotension (Vascular disorders) | 11 (11)
Dizziness (Nervous system disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortezomib and Dexamethasone (N=35)
alkaline phosphatase elevated (Investigations) | 4 (4)
drug rash (Blood and lymphatic system disorders) | 3 (3)
tinnitus (Ear and labyrinth disorders) | 2 (2)
nausea (Gastrointestinal disorders) | 15 (15)
diarrhea (Gastrointestinal disorders) | 14 (14)
adrenal insufficiency (Endocrine disorders) | 4 (4)
constipation (Gastrointestinal disorders) | 13 (13)
anorexia (Gastrointestinal disorders) | 5 (5)
abdominal distension (Gastrointestinal disorders) | 4 (4)
hypotension (Vascular disorders) | 8 (8)
alopecia (Skin and subcutaneous tissue disorders) | 14 (14)
rash (Skin and subcutaneous tissue disorders) | 7 (7)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (10)
sinus tachycardia (Cardiac disorders) | 16 (16)
muscle weakness (Musculoskeletal and connective tissue disorders) | 5 (5)
dizziness (Nervous system disorders) | 4 (6)
anxiety (Nervous system disorders) | 7 (12)
Blurred vision (Eye disorders) | 7 (7)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 12 (14)
cough (Respiratory, thoracic and mediastinal disorders) | 6 (7)
peripheral edema (General disorders) | 5 (5)
petechiae (Blood and lymphatic system disorders) | 4 (4)
oral mucositis (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes